CLINICAL TRIAL: NCT01545388
Title: A Phase III, Randomized, Placebo and Active-Controlled, Double-Blind Clinical Trial to Study the Efficacy and Safety of the Addition of Metformin in Japanese Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Diet/Exercise Therapy and Sitagliptin Monotherapy
Brief Title: Metformin Add-on Regimen Comparison Study in Japanese Participants With Type 2 Diabetes Mellitus (MK-0431A-136)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431A-136; ONO-5435A (Other: ONO Pharmaceutical Company, Ltd.)
Record Dates: First submitted 2012-03-01; First posted 2012-03-06 (Estimated); Results first posted 2014-03-26 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Metformin 500 mg q.d. (Experimental): Participants will receive sitagliptin daily (continuing their pre-study dose), 2 metformin 250 mg tablets in the morning and 1 matching placebo tablet in the evening.
  Interventions: Drug: Sitagliptin; Drug: Metformin; Drug: Placebo
- Metformin 250 mg b.i.d. (Experimental): Participants will receive sitagliptin daily (continuing their pre-study dose), 1 metformin 250 mg tablet and 1 matching placebo tablet in the morning and 1 metformin 250 mg tablet in the evening.
  Interventions: Drug: Sitagliptin; Drug: Metformin; Drug: Placebo
- Placebo (Placebo Comparator): Participants will receive sitagliptin daily (continuing their pre-study dose), 2 matching placebo tablets in the morning and 1 matching placebo tablet in the evening.
  Interventions: Drug: Sitagliptin; Drug: Placebo

INTERVENTIONS:
Drug: Sitagliptin — Sitagliptin, orally, 50 or 100 mg tablet (continuation of the pre-study dose)
  Other Names: MK-0431/ONO-5435
Drug: Metformin — Metformin, orally, 500 mg daily (single dose; two 250 mg tablets) for 24 weeks
  Arms: Metformin 500 mg q.d.
Drug: Metformin — Metformin, orally, 500 mg daily (divided dose; 250 mg tablet b.i.d.) for 24 weeks
  Arms: Metformin 250 mg b.i.d.
Drug: Placebo — Placebo to match metformin 250 mg tablets, orally, for 24 weeks

SUMMARY:
This study will evaluate the effect of the addition of metformin once daily (q.d.) or twice daily (b.i.d.) to sitagliptin monotherapy in Japanese participants with Type 2 diabetes mellitus (T2DM) who have inadequate glycemic control with diet/exercise therapy and sitagliptin monotherapy. The primary hypotheses are that the addition of metformin 250 mg b.i.d. or metformin 500 mg q.d. is superior to the addition of placebo on the change from baseline in hemoglobin A1c (HbA1c) at 24 weeks and that the addition of metformin 500 mg q.d. is non-inferior to the addition of metformin 250 mg b.i.d. on the change from baseline in HbA1c at 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus (T2DM)
* Currently being treated with diet/exercise and on stable dose of sitagliptin for ≥ 4 weeks, on any additional oral hypoglycemic agent (AHA) in the prior 8 weeks, and HbA1c ≥ 6.0% and ≤ 9.0%; or
* Currently being treated with diet/exercise and on stable dose of sitagliptin for ≥ 10 weeks, not on any additional oral AHA in the prior 8 weeks, and HbA1c ≥ 6.5% and < 10.0%

Exclusion Criteria:

* Type 1 diabetes mellitus,
* Secondary diabetes mellitus, or
* Gestational diabetes mellitus

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2012-02-23 (Actual); Primary Completion 2013-03-12 (Actual); Study Completion 2013-03-12 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0431A-136&kw=0431A-136&tab=access

RESULTS

PARTICIPANT FLOW:
Groups:
- Metformin 500 mg q.d.: Participants received sitagliptin daily at pre-study dose, 2 metformin 250 mg tablets in the morning and 1 matching placebo tablet in the evening.
- Metformin 250 mg b.i.d.: Participants received sitagliptin daily at pre-study dose, 1 metformin 250 mg tablet and 1 matching placebo tablet in the morning and 1 metformin 250 mg tablet in the evening.
- Placebo: Participants received sitagliptin daily at pre-study dose, 2 matching placebo tablets in the morning and 1 matching placebo tablet in the evening.
Period: Overall Study
Arm/Group | Metformin 500 mg q.d. | Metformin 250 mg b.i.d. | Placebo
Started | 138 | 133 | 66
Completed | 130 | 122 | 58
Not Completed | 8 | 11 | 8
Not completed — Adverse Event | 2 | 4 | 1
Not completed — Lack of Efficacy | 3 | 2 | 5
Not completed — Participant moved or relocated | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 4 | 2
Not completed — Other | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants as treated population defined as all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin 500 mg q.d. | Metformin 250 mg b.i.d. | Placebo | Total
Number analyzed (Participants) | 138 | 133 | 66 | 337
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.46 (9.61) | 59.65 (9.22) | 60.05 (9.30) | 59.65 (9.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 46 | 28 | 126
  Male | 86 | 87 | 38 | 211
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percent of glycosylated hemoglobin] | 7.60 (0.83) | 7.40 (0.68) | 7.53 (0.77) | 7.51 (0.76)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] | 158.58 (32.45) | 148.98 (26.27) | 154.27 (27.51) | 153.95 (29.42)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 24 in Hemoglobin A1c (HbA1c)
Description: Based on a constrained longitudinal data analysis (cLDA) model with terms for treatment, other prior antihyperglycemic agent (AHA) therapy status other than sitagliptin (yes/no), study drug regimen (just before meal/after meal), sitagliptin dosage (50 mg/100 mg), time and the interaction of time by treatment, time by other prior AHA therapy status, time by study drug regimen, time by sitagliptin dosage and study drug regimen by sitagliptin dosage, with a constraint that the mean baseline is the same for all treatment groups.
Time Frame: Baseline and Week 24
Population: Per-protocol population defined as all randomized participants who had at least one measurement (baseline or post-randomization), with participants and/or selected data excluded due to protocol violations.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent of glycosylated hemoglobin
Arm/Group | Metformin 500 mg q.d. | Metformin 250 mg b.i.d. | Placebo
Number analyzed (Participants) | 136 | 130 | 66
Percent of glycosylated hemoglobin | -0.434 [-0.553 to -0.315] | -0.587 [-0.708 to -0.467] | 0.091 [-0.073 to 0.255]
Statistical Analysis 1: Comparison: Metformin 250 mg b.i.d. vs Placebo; Test type: Superiority or Other; p < 0.001, cLDA; Based on a cLDA model with the terms listed above and a constraint that the mean baseline is the same for all treatment groups; Difference in least squares means = -0.678, 95% CI 2-sided [-0.868 to -0.489]
Statistical Analysis 2: Comparison: Metformin 500 mg q.d. vs Placebo; Test type: Superiority or Other; p < 0.001, cLDA; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = -0.525, 95% CI 2-sided [-0.713 to -0.337]
Statistical Analysis 3: Comparison: Metformin 500 mg q.d. vs Metformin 250 mg b.i.d; Test type: Non-Inferiority or Equivalence — The non-inferiority margin (Δ) is set as 0.3% to show the non-inferiority of metformin 500 mg q.d. to metformin 250 mg b.i.d; Difference in least squares means = 0.153, 95% CI 2-sided [0.000 to 0.306]

2. Secondary Outcome: Change From Baseline to Week 24 in Fasting Plasma Glucose (FPG)
Description: Based on a cLDA model with terms for treatment, other prior AHA therapy status other than sitagliptin (yes/no), study drug regimen (just before meal/after meal), sitagliptin dosage (50 mg/100 mg), time and the interaction of time by treatment, time by other prior AHA therapy status, time by study drug regimen, time by sitagliptin dosage and study drug regimen by sitagliptin dosage, with a constraint that the mean baseline is the same for all treatment groups.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Metformin 500 mg q.d. | Metformin 250 mg b.i.d. | Placebo
Number analyzed (Participants) | 136 | 130 | 66
mg/dL | -9.02 [-13.74 to -4.30] | -11.27 [-16.07 to -6.46] | 7.32 [0.86 to 13.79]
Statistical Analysis 1: Comparison: Metformin 250 mg b.i.d. vs Placebo; Test type: Superiority or Other; p < 0.001, cLDA; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = -18.59, 95% CI 2-sided [-25.94 to -11.24]
Statistical Analysis 2: Comparison: Metformin 500 mg q.d. vs Placebo; Test type: Superiority or Other; p < 0.001, cLDA; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = -16.34, 95% CI 2-sided [-23.62 to -9.06]
Statistical Analysis 3: Comparison: Metformin 500 mg q.d. vs Metformin 250 mg b.i.d; Test type: Superiority or Other; Difference in least squares mean = 2.25, 95% CI 2-sided [-3.63 to 8.14]

3. Primary Outcome: Percentage of Participants Who Experienced at Least One Adverse Event
Time Frame: Up to 26 weeks
Population: All participants as treated defined as all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Metformin 500 mg q.d. | Metformin 250 mg b.i.d. | Placebo
Number analyzed (Participants) | 138 | 133 | 66
Percentage of participants | 65.9 | 67.7 | 60.6

4. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to an Adverse Event
Time Frame: Up to 24 weeks
Population: All participants as treated defined as all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Metformin 500 mg q.d. | Metformin 250 mg b.i.d. | Placebo
Number analyzed (Participants) | 138 | 133 | 66
Participants | 2 | 3 | 1

ADVERSE EVENTS:
Time Frame: Up to 26 weeks
Description: All participants as treated defined as all randomized participants who received at least one dose of study treatment.
Arm/Group | Metformin 500 mg q.d. | Metformin 250 mg b.i.d. | Placebo
Serious Adverse Events (participants affected / at risk) | 4/138 | 2/133 | 0/66
Other Adverse Events (participants affected / at risk) | 29/138 | 35/133 | 8/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin 500 mg q.d. (N=138) | Metformin 250 mg b.i.d. (N=133) | Placebo (N=66)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Brain stem infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin 500 mg q.d. (N=138) | Metformin 250 mg b.i.d. (N=133) | Placebo (N=66)
Constipation (Gastrointestinal disorders) | 8 (8) | 5 (6) | 0 (0)
Nasopharyngitis (Infections and infestations) | 17 (21) | 28 (31) | 7 (7)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 4 (5) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation.

Any information identified by the sponsor as confidential must be deleted prior to submission.